CLINICAL TRIAL: NCT02840175
Title: Treatment Tapering in Oligoarticular or Rheumatoid Factor Negative Polyarticular Juvenile Idiopathic Arthritis With Inactive Disease on Biologic Therapy
Brief Title: Treatment Tapering in JIA With Inactive Disease
Acronym: AJIBIOREM
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: P 150902; 2016-000312-15 (EudraCT Number)
Record Dates: First submitted 2016-07-19; First posted 2016-07-21 (Estimated); Last update posted 2021-04-01 (Actual); Status verified 2021-03

CONDITIONS: Juvenile Idiopathic Arthritis
Keywords: Treatment tapering; Oligoarticular; Juvenile Idiopathic Arthritis; Inactive disease; Biologic therapy
MeSH Terms: conditions — Arthritis, Juvenile | interventions — Etanercept; Adalimumab; Abatacept; tocilizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): * Day 0 at Weeks 24 : Increase the interval between 2 doses of the biological agent (etanercept, adalimumab, tocilizumab, abatacept)
  * Weeks 24 at Weeks 72: Stop the biological agent if inactive disease is maintained.
  Interventions: Drug: etanercept; Drug: adalimumab; Drug: Abatacept; Drug: Tocilizumab
- Control (Active Comparator): * Day 0 at Weeks 24: Maintain the biological agent (etanercept, adalimumab, tocilizumab, abatacept) at the same dose.
  * Weeks 24 at Weeks 48 : Increase the interval between 2 doses of the biological agent.
  * Weeks 48 at Weeks 72: Stop the biological agent if inactive disease is maintained.
  Interventions: Drug: etanercept; Drug: adalimumab; Drug: Abatacept; Drug: Tocilizumab

INTERVENTIONS:
Drug: etanercept — will be tapered from every week to every 2 weeks for 12 weeks then to every 3 weeks for 12 weeks
  Other Names: Enbrel®
Drug: adalimumab — will be tapered from every 2 weeks to every 3 weeks for 12 weeks and to every 4 weeks for 12 weeks
  Other Names: Humira®
Drug: Abatacept — will be tapered from every 4 weeks to every 6 weeks for 24 weeks
  Other Names: Orencia®
Drug: Tocilizumab — will be tapered from every 4 weeks to every 6 weeks for 24 weeks
  Other Names: RoActemra®

SUMMARY:
As biologic treatments are expensive and associated with some concerns regarding long-term safety, investigator hypothesize that early tapering and then withdrawal of biological agent, in an homogenous group of children with juvenile idiopathic arthritis achieving inactive disease, is safe and not inferior to the maintenance of stable treatment intensity over 24 weeks. In addition, investigator also hypothesize that an earlier tapering of treatment is associated with a better quality-of-life and a general cost saving effect. MRP8/14 will be studied as a potential biomarker for the risk of relapse. A study for biologic agent, anti-biologic agent antibodies and a pharmacogenomic approach will complete the research, as pharmacokinetic study during withdrawal of biologic treatment are rare in children.

DETAILED DESCRIPTION:
Juvenile idiopathic arthritis (JIA) is characterized by chronic arthritis of unknown etiology starting before the age of 16. There are four to five thousand paediatric patients with JIA in France. Most of these patients are diagnosed with oligoarticular or rheumatoid factor negative polyarticular JIA. The prognosis of the disease has dramatically improved thanks to the introduction of biologic agents in patients with an extended oligoarticular or rheumatoid factor negative polyarticular JIA and inadequate response to methotrexate. Inactive disease and long-lasting clinical remission are achieved in most cases. "Treat to target" approaches are increasingly recommended, with earlier introduction of biologics, however the way to taper or withdraw treatment in patients achieving inactive disease is not codified. As biologic treatments are expensive and associated with some concerns regarding long-term safety, this study aim to test, in a randomized fashion, the hypothesis that early tapering of biologic agents (i.e. increasing the intervals between injections as soon as inactive disease is documented) is safe and non-inferior to the maintenance of stable treatment intensity over 24 weeks, and therefore test the possibility of early biologic agent withdrawal. It will also study concentrations of different biological agent, the occurrence of anti-drugs antibodies while tapering and then withdrawing biologics, and their possible association with a higher risk of relapse. In addition, investigators will test if the serum level of proteins 100 (MRP8/14) could be predictive of flares. Finally, pharmaco-economic analyses and quality of life studies will be conducted.

ELIGIBILITY:
Inclusion Criteria:

* Patient aged 2 to 17 years and treated with etanercept or tocilizumab or adalimumab, or patient aged 6 to 17 years and treated with abatacept.
* Patient with an oligoarticular or polyarticular rheumatoid factor negative JIA
* Patient treated with biologic treatment for persistent arthritis according to the marketing authorization.
* Patient who achieved inactive disease within two years of treatment with the last biologic agent administered, according to Wallace criteria : no joints with active arthritis, no active uveitis (as defined by the SUN Working Group), ESR or CRP level within normal limits in the laboratory where tested (or, if elevated, not attributable to JIA), physician's global assessment of disease activity score (< 10/100 visual analogue scale), and duration of morning stiffness < ou = 15 minutes (within 7 days before the visit).
* Patient with inactive disease achieved for less than 12 months.
* Patient with stable doses of non-steroidal anti-inflammatory drugs, Methotrexate (maximum 20 mg/m2/week), and other non biologic DMARD for at least one month before inclusion
* Patient without steroids or joint injection or live vaccines injection for at least one month.
* Signed informed consent by both parents (or legal guardian) and patient's agreement.
* Patient affiliated to the National Health Assurance system.

Exclusion Criteria:

* Patient with systemic form, rheumatoid factor positive, psoriatic or associated with enthesitis related JIA.
* Patient undergoing biologic therapy due to JIA-associated uveitis or with active uveitis at time of randomization.
* Patient with any contraindication to continue ongoing biologic treatment, notably ongoing uncontrolled infection, suspicion or evidence of demyelinating disease of the central nervous system.
* Patient previously treated with the same biotherapy for which dose decreasing or biotherapy withdrawal was already tested in the past for inactive disease and then reintroduced.
* Pregnancy or absence of effective contraception (including abstinence) in a pubertal patient.
* Patient suffering from tuberculosis.
* Patient with moderate to severe cardiac failure (NYHA class III / IV).

Ages: 2 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 62 (Actual)
Dates: Start 2017-05-18 (Actual); Primary Completion 2019-10-29 (Actual); Study Completion 2020-10-01 (Actual)

PRIMARY OUTCOMES:
Persistence of inactive disease | 24 weeks
  Inactive disease is defined by the criterion of Wallace :
  * No joints with active arthritis,
  * No active uveitis as defined by the SUN Working Group2 (The Standardization of Uveitis Nomenclature (SUN) Working Group defines inactive anterior uveitis as "grade zero cells," indicating <1 cell in field sizes of 1 mm by a 1-mm slit beam),
  * Erythrocyte sedimentation rate (ESR) ≤ 20 mm or C-reactive protein (CRP) level ≤ 10 mg/L (or ≤ 1 mg/dl or ≤ 100 µg/dl) or, if elevated, not attributable to JIA (if both ESR and CRP are available, both of them should be in the normal range)
  * Physician's global assessment of disease activity score (< 10/100 visual analogue scale),
  * and duration of morning stiffness < or egal to 15 minutes (within 7 days before the visit).
  For all the visits, joint counts and physician global assessment of disease activity will be performed by an investigator blinded from patient study group.

SECONDARY OUTCOMES:
Adverse and serious adverse events or of special interest | Weeks 12, 24, 36, 48, 60, 72
Persistent inactive disease as defined by Wallace criteria | 72 weeks
Juvenile Arthritis Disease Activity Score (JADA score) | Day 0, Weeks 12, 24, 48, 72
Biological agent concentrations | Day 0, weeks 12, 24, 36, 48, 60
  according to drug administration (Etanercept or Abatacept or Tocilizumab or Adalimumab)
Anti-drugs antibodies concentrations | Day 0, weeks 12, 24, 36, 48, 60
  anti-Etanercept or anti-Abatacept or anti-Tocilizumab or anti-Adalimumab
Proteins S100 concentrations (MRP8/14 level) | Day 0, weeks 24, 48, 72
Concentration of additional informative markers (cytokines, chemokines) | Day 0, weeks 24, 48, 72
score of quality of life with the Paediatric Quality of Life (PedsQL) | Day 0, weeks 24, 36, 72
score of quality of life with the Childhood Health Assessment Questionnaire (CHAQ) | Day 0, weeks 12, 24, 36, 72
score of quality of life with the Life Quality Questionnaire related to the health (EQ-5D Y) | Day 0, weeks 24, 36, 72
cost of early treatment tapering and withdrawal | weeks 12, 24, 36, 60, 72
cost of late treatment tapering and withdrawal | weeks 12, 24, 36, 60, 72

CONTACTS AND LOCATIONS:
Overall Officials: Florence UETTWILLER, PhD, Study Chair — Necker Children's Hospital, Paris, France
Locations (1):
- Necker Children's Hospital, Paris, France

IPD SHARING:
Plan to Share IPD: No